CLINICAL TRIAL: NCT03982147
Title: White Matter Connections and Memory: the STRATEGIC Study
Acronym: STRATEGIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Mike O'Sullivan, Chief Investigator, King's College London
Other Study IDs: KCH14-072; 13/LO/1745 (Other: London Bromley Research Ethics Committee); K022113 (Other Grant/Funding Number: Medical Research Council, UK)
Record Dates: First submitted 2018-11-23; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Stroke; Cognitive Impairment; Memory Impairment
Keywords: Diffusion tensor imaging
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Patients with recent ischaemic stroke

SUMMARY:
In patients who have had a stroke, memory problems are common. Some patients with memory problems improve over the first year after stroke, but recovery is unpredictable. The STRATEGIC study assesses patients with recent stroke and follows them up after one year. The study uses cognitive testing and advanced MRI to understand the brain's mechanism for recovery from memory problems and to identify factors that may predict later recovery.

DETAILED DESCRIPTION:
Memory breakdown in older age is a major challenge for medical research, with an increasing burden in personal, societal and fiscal terms. Stroke is an important cause. Memory depends on widespread networks in the brain which are bound together by white matter connections, which essentially act as the wiring of brain networks. This project uses a technique called diffusion tensor MRI to investigate these connections and their relationship to brain function and patterns of memory impairment after stroke.

Previous research showed that a tract called the fornix was most important in the healthy brain and in ageing. However, in individuals at an early stage of memory decline alternative pathways became disproportionately more important. This led to the idea that individuals with early memory decline might be especially vulnerable to injury to these alternative tracts from stroke. The purpose of this project is to test this idea.

The project focuses on patients with recent stroke. Participants undergo MRI, including diffusion tensor MRI, and in-depth testing of memory and other cognitive functions. The pattern of damage to temporal lobe connections in the brain will be assessed and related to the impact of brain infarction on memory. Analysis will determine how undamaged tracts contribute to recovery over one year. Finally, cutting edge computational image analysis techniques will be applied to try and predict memory profile in more detail and extract maximum information about prognosis from brain images.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 50 years
* Recent ischaemic stroke
* English is first language

Exclusion Criteria:

* Previous large artery infarct
* Major neurological or psychiatric condition
* Moderate to severe head injury (Mayo classification)
* Dementia
* Severe cardiac failure
* Active malignancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent ischaemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score at 30-90 days | 30-90 days after stroke
  The MoCA is a widely used test measuring across several cognitive domains. It gives a score out of 30.
  https://www.mocatest.org
Montreal Cognitive Assessment (MoCA) score at one year | One year after stroke
  The MoCA is a widely used test measuring across several cognitive domains. It gives a score out of 30.
  https://www.mocatest.org
Montreal Cognitive Assessment (MoCA), change in score over one year | From 30-90 days after stroke to one year after stroke
  The MoCA is a widely used test measuring across several cognitive domains. It gives a score out of 30.
  https://www.mocatest.org
Verbal free recall score on the Free and Cued Selective Reminding Task (FSCRT) at 30-90 days | 30-90 days after stroke
  The FCSRT tests how well participants can remember 16 words. Participants make three attempts, giving a total score out of 48. The test has been widely used in studies of memory and is described in Grober, E., & Buschke, H. (1987). Genuine memory deficits in dementia. Developmental Neuropsychology, 3, 13-36.
Verbal free recall score on the Free and Cued Selective Reminding Task (FSCRT) at one year | One year after stroke
  The FCSRT tests how well participants can remember 16 words. Participants make three attempts, giving a total score out of 48. The test has been widely used in studies of memory and is described in Grober, E., & Buschke, H. (1987). Genuine memory deficits in dementia. Developmental Neuropsychology, 3, 13-36.
Verbal free recall score on the Free and Cued Selective Reminding Task (FSCRT), change in score over one year | From 30-90 days after stroke to one year after stroke
  The FCSRT tests how well participants can remember 16 words. Participants make three attempts, giving a total score out of 48. The test has been widely used in studies of memory and is described in Grober, E., & Buschke, H. (1987). Genuine memory deficits in dementia. Developmental Neuropsychology, 3, 13-36.
Backward digit span score at 30-90 days | 30-90 days after stroke.
  The digit span test measures working memory and is taken from the Wechsler Adult Intelligence Scale IV. In the test participants must repeat a sequence of digits. Sequences are repeated at increasing length until the participant makes two errors at the same length. The test comprises two parts. In the first, participants repeat sequences is the order given; in the second they repeat sequences in reverse order. This outcome measure takes the total correct responses in reverse order. Sequence lengths are between two and seven digits, with to sequences of each length, giving a maximum score of 12.
Backward digit span score at one year | One year after stroke
  The digit span test measures working memory and is taken from the Wechsler Adult Intelligence Scale IV. In the test participants must repeat a sequence of digits. Sequences are repeated at increasing length until the participant makes two errors at the same length. The test comprises two parts. In the first, participants repeat sequences is the order given; in the second they repeat sequences in reverse order. This outcome measure takes the total correct responses in reverse order. Sequence lengths are between two and seven digits, with to sequences of each length, giving a maximum score of 12.
Backward digit span score, change in score over one year | From 30-90 days after stroke to one year after stroke
  The digit span test measures working memory and is taken from the Wechsler Adult Intelligence Scale IV. In the test participants must repeat a sequence of digits. Sequences are repeated at increasing length until the participant makes two errors at the same length. The test comprises two parts. In the first, participants repeat sequences is the order given; in the second they repeat sequences in reverse order. This outcome measure takes the total correct responses in reverse order. Sequence lengths are between two and seven digits, with to sequences of each length, giving a maximum score of 12.
Paired Associate Learning (PAL) recognition score at 30-90 days | 30-90 days after stroke.
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recognition score is the number of correct choices when given two possible locations for a given object. Each object is tested three times, giving a maximum score of 30.
Paired Associate Learning (PAL) recognition score at one year | One year after stroke.
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recognition score is the number of correct choices when given two possible locations for a given object. Each object is tested three times, giving a maximum score of 30.
Paired Associate Learning (PAL) recognition score, change in score over one year | From 30-90 days after stroke to one year after stroke
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recognition score is the number of correct choices when given two possible locations for a given object. Each object is tested three times, giving a maximum score of 30.
Paired Associate Learning (PAL) recall score at 30-90 days | 30-90 days after stroke
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recall score measures participants ability to recall which object was present at each location (a maximum of 10).
Paired Associate Learning (PAL) recall score at one year | One year after stroke
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recall score measures participants ability to recall which object was present at each location (a maximum of 10).
Paired Associate Learning (PAL) recall score, change in score over one year | From 30-90 days after stroke to one year after stroke
  The PAL task measures participants' ability to associate two items of information in memory. In this study, participants must learn a set of ten objects and their associated locations. The recall score measures participants ability to recall which object was present at each location (a maximum of 10).
Process Dissociation Procedure (PDP) familiarity score at 30-90 days | 30-90 days after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.
Process Dissociation Procedure (PDP) familiarity score at one year | One year after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.
Process Dissociation Procedure (PDP) familiarity score, change in score over one year | From 30-90 days after stroke to one year after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.
Process Dissociation Procedure (PDP) recollection score at 30-90 days | 30-90 days after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.
Process Dissociation Procedure (PDP) recollection score at one year | One year after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.
Process Dissociation Procedure (PDP) recollection score, change in score over one year | From 30-90 days after stroke to one year after stroke
  The PDP is a word memory test. Participants first read out loud a set of words. They are then presented with incomplete words and must fill in the missing letters. In one part of the test, participants must use one of the remembered words whenever possible. In the other part of the test, they must avoid the remembered words. The two parts are designed to dissociate two types of memory: familiarity and recollection. Familiarity is the unconscious remembering of a word because it was previously seen, which is an advantage when including the words, but a disadvantage when avoiding them. Recollection is the conscious remembering of a word and the context where it was encountered. This is an advantage in both parts of the test. The scores in each part of the test are combined to compute scores for familiarity and recollection, each in percent.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J O'Sullivan, MBBS,PhD, Principal Investigator — King's College London and University of Queensland

IPD SHARING:
Plan to Share IPD: Undecided
If possible, we hope to share anonymised test scores and derived MRI measures, along with demographic and other background data.